CLINICAL TRIAL: NCT06677125
Title: Magnetic Mallet Versus Densah Bur for Crestal Sinus Left With Implant Placement in Maxilla (Randomized Controlled Clinical Trial)
Brief Title: Magnetic Mallet and Densah Bur for Crestal Sinus Left
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 814-12
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Maxillary Sinus Left

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Procedure: Electrical Mallet
- Control Group (Active Comparator)
  Interventions: Procedure: Densah bur

INTERVENTIONS:
Procedure: Electrical Mallet — The osteotome will be directly attached and pushed by magnetic mallet and a shock wave will be pushed on their tip. The electrical mallet will be imparted to osteotomes a longitudinal movement along a central axis moving up and down toward pilot bone hole providing a driving mechanism of longitudinal movements. Then the sinus lift instruments (Sweden and Martina) will be used to slowly lift the sinus. After that implant will be placed with the help of implant drilling device.
  Arms: Test Group
Procedure: Densah bur — The implant motor will be adjusted on reverse-densifying mode with 800 to 1200 rpm. According to the desired implant dimension, it will be started with the smallest densah bur. The first densah bur will advanced in densifying mode with bouncing motion in and out movement with copious irrigation until.
  Arms: Control Group

SUMMARY:
Background: Implant placement in the posterior maxilla is problematic procedure, not only due to inferior properties of bone but also due to loss of vertical bone height, which happens after extraction of posterior teeth. When the required additional height is few millimeters, indirect transcrestal sinus lifting is recommended. Aim: The aim of this study is to evaluate Densah bur versus Magnetic mallet in transcrestal sinus lifting procedure in edentulous molar and premolar maxillary region.

ELIGIBILITY:
Inclusion Criteria:

* Patient seeking replacement of missing maxillary posterior teeth by dental implant procedure.
* Residual bone height is (5-7) mm measured from crestal bone to sinus floor.
* Both genders.
* Good general health;
* Good oral hygiene.

Exclusion Criteria:

* Uncontrolled Diabetes.
* Coagulation disorders.
* Immunological disorders.
* Previous radiation of the head and neck region.
* Presence of chronic systemic diseases;
* Presence of acute or chronic sinus problems;
* Alcohol or drug abuse;
* Heavy smokers.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain socres | 3rd day, 1 week and 10 days
  pain will be examined using visual analogue scale (VAS) 0 means no pain 10 means extreme pain
change in implant stability | baseline and 4 months
  will be measured by the Resonance Frequency Analysis using osstel

SECONDARY OUTCOMES:
change in implant protrusion length | baseline and 4 months
  Immediate post- operative CBCT (T1) will be done to measure the implant protrusion length (IPL) which is the length of the implant extending into the maxillary sinus.
change in bone density | baseline and 4 months
  it will be measured by CBCT
change in prescence of complications | 3rd day, 1 week and 10 days
  patients will be followed up to assess the occurence of any clincial complications

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt